CLINICAL TRIAL: NCT03633097
Title: Efficacy and Safety of Acupuncture Treatment as an Adjunctive Therapy After Knee Replacement - Single-center, Pragmatic, Randomized, Assessor Blinded, Pilot Study-
Brief Title: Efficacy and Safety of Acupuncture Treatment as an Adjunctive Therapy After Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Oriental Medical Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Yun-Kyung Song, Sponsor-principle investigator, Gachon University Gil Oriental Medical Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISEE_2018_TKA_A
Record Dates: First submitted 2018-07-31; First posted 2018-08-16 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Knee Replacement; Acupuncture
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single blinded, outcome assessor blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture + Usual care (Experimental): Acupuncture with Cnoxane Injection 40mg, Esomezol Capsule, Synerjet Semi Tablet and Ocoron Tablet
  Interventions: Other: Acupuncture and Usual care
- Usual care (Active Comparator): Cnoxane Injection 40mg, Esomezol Capsule, Synerjet Semi Tablet and Ocoron Tablet
  Interventions: Drug: Usual care

INTERVENTIONS:
Other: Acupuncture and Usual care — patients after surgery receive usual care(Cnoxane Injection 40mg, Esomezol Capsule, Synerjet Semi Tablet and Ocoron Tablet) as well as acupuncture treatment as an adjunctive therapy
  Arms: Acupuncture + Usual care
Drug: Usual care — patients after surgery receive usual care alone(Cnoxane Injection 40mg, Esomezol Capsule, Synerjet Semi Tablet and Ocoron Tablet)
  Arms: Usual care

SUMMARY:
Efficacy and Safety of Acupuncture Treatment as an Adjunctive Therapy After Knee Replacement

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of osteoarthritis and listed for an unilateral total knee replacement.
* Subject has a normal cognitive function
* Subject is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Those who have undergone total knee arthroplasty due to gout
* Those who have had total knee arthroplasty due to trauma
* Those who have had total knee arthroplasty due to autoimmune related diseases such as rheumatoid arthritis
* Those who are participating in other clinical trials
* Those who have a history of participating in other clinical trials within one month
* Those who are difficult to write a research consent form
* Those who are judged to be inappropriate for the clinical study by the researchers.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Korean version of Western Ontario and McMaster Universities Arthritis Index | Screening, day 11, day 21
  K-WOMAC is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales

SECONDARY OUTCOMES:
Change from baseline in Numeric rating scale | Screening, baseline, day 5, 11, 21, 28, 84
  NRS range was 0-10 with 0 being no pain and 10 the worst pain possible.
Change from baseline in Physical Condition related with mobility at every visit | Screening, day 11, day 84
  mobility (5 meters walking test at comfortable speed - 5mWT) (meters/second)
Change from baseline in Physical Condition related with endurance at every visit | Screening, day 11, day 84
  endurance (Sit-to-stand test - STS) (seconds)
Change from baseline in Timed Up and Go Test at every visit | Screening, day 11, day 84
  a functional test evaluating the time to rise from a chair, walk 3 meters, turn around, walk back to the chair and sit down (abnormal cut-off value >12 seconds).
Change from baseline in Alternative-Step Test at every visit | Screening, day 11, day 84
  a functional test measuring clinical balance performance, and it has been shown to predict fall risk among elderly subjects (seconds)
Change from baseline in Range of motion | Screening, baseline, day 5, 11, 28, 84
  Compare flexion and extension angle using long arm goniometer between experimental and comparator group

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kyung Song, PhD, Principal Investigator — Gachon university of Gil oriental hospital
Locations (2):
- South Korea (2):
  - Catholic Kwandong University International St. Mary'S Hospital, Incheon
  - Catholic Kwandong University International St. Mary'S Hospita, Incheon

REFERENCES:
- [Derived] Park TY, Kim HJ, Lee JH, Sunwoo YY, Do KS, Han SN, Song YK, Chae DS. Efficacy and safety of acupuncture treatment as an adjunctive therapy after knee replacement: Single-center, pragmatic, randomized, assessor blinded, pilot study. Medicine (Baltimore). 2021 Mar 12;100(10):e24941. doi: 10.1097/MD.0000000000024941. PMID 33725856